CLINICAL TRIAL: NCT04818060
Title: Preparing for Prevention of Huntington's Disease (PREVENT-HD)
Acronym: PREVENT-HD
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-1175; A535100 (Other: UW Madison); SMPH/NEUROLOGY/NEUROLOGY (Other: UW Madison); Protocol Version 7/17/2024 (Other: UW Madison); 7U01NS105509 (NIH); 7U01NS103475 (NIH)
Record Dates: First submitted 2021-03-15; First posted 2021-03-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Huntington Disease
Keywords: biomarkers; premanifest HD; early diagnosis; motor impairment
MeSH Terms: conditions — Huntington Disease; Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebral spinal fluid (22mL) and blood samples (two tubes, 20mL each).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low Risk of Motor Diagnosis: Approximately 52 participants who have a low probability of motor diagnosis based on the multivariate risk score.
  Interventions: Other: Clinical Assessments; Diagnostic Test: MRI Scan; Diagnostic Test: Lumber Puncture (LP)
- High Risk of Motor Diagnosis: Approximately 102 participants who have a high probability of motor diagnosis based on the multivariate risk score.
  Interventions: Other: Clinical Assessments; Diagnostic Test: MRI Scan; Diagnostic Test: Lumber Puncture (LP)
- Stage I or II Huntington's Disease: Approximately 52 participants who are living with diagnosed stage I or stage II Huntington's Disease.
  Interventions: Other: Clinical Assessments; Diagnostic Test: MRI Scan; Diagnostic Test: Lumber Puncture (LP)
- Healthy Controls: Approximately 52 participants who are age-, ethnicity-, and education-matched healthy controls.
  Interventions: Other: Clinical Assessments; Diagnostic Test: MRI Scan; Diagnostic Test: Lumber Puncture (LP)

INTERVENTIONS:
Other: Clinical Assessments — A neurological evaluation will be administered to all participants at baseline, 1 year and 2 year follow-up visits. Motor exams and premorbid IQ assessments will be video-recorded for rater reliability assessments conducted randomly throughout the research project.
Diagnostic Test: MRI Scan — At baseline and 2 year follow-up all participants will undergo a 60-minute 3T MRI scanning session which will consist of measures of the volume of brain tissue and cerebral spinal fluid, as well as connections in the brain measuring water pathways and pictures of the brain active and at rest.
Diagnostic Test: Lumber Puncture (LP) — Participants will be asked to complete a LP at both onsite study visits (baseline and 2 year follow-up). Blood collection following the procedure will consist of about 80mL and will be stored at a repository for biomarker analysis.

SUMMARY:
This is a prospective investigation which aims to address key challenges to the design of clinical trials to prevent the onset of Huntington's disease (HD). The project will provide necessary psychometric data for clinical outcome assessments (COAs) and biomarkers (BMs) in the cerebral spinal fluid (CSF) to address questions of central importance to the success of these measures for premanifest clinical trials. Of the 258 participants: 52 will be low risk of motor diagnosis, 102 high risk of motor diagnosis, 52 with diagnosed HD (stages I or II), and 52 healthy controls. Participants can expect to be in the study for up to 2 years.

DETAILED DESCRIPTION:
This is a prospective investigation which aims to address key challenges to the design of clinical trials to prevent the onset of Huntington's disease (HD). The project will provide necessary psychometric data for clinical outcome assessments (COAs) and biomarkers (BMs) in the cerebral spinal fluid (CSF) to address questions of central importance to the success of this measure for premanifest clinical trials such as:

1. How reliable the measure is in the same person when repeated over time;
2. how reliable the measure is in the same person when analyzed by two different labs/sites;
3. how well the measure reflects disease symptoms;
4. how well the measure predicts meaningful disease outcomes;
5. how well the measure tracks disease progression or severity; AND
6. how many research subjects are required to test that an intervention is delaying/slowing the onset of HD?

Answers to these questions will better position the field to more effectively test new interventions to prevent HD such as gene therapies and new drugs.

Neurocognitive, motor and behavioral data, blood, CSF, and genetic samples, and MRI measures will be collected from 258 participants at baseline. Of the 258 participants: 52 will be low risk of motor diagnosis, 102 high risk of motor diagnosis, 52 with diagnosed HD (stages I or II), and 52 healthy controls. Neurocognitive and behavioral data, blood and CSF samples, and MRI will be repeated 2 years (18-24 months) after the baseline visit. Remote assessments of clinical outcome measures (neurocognitive, motor and behavioral data) will be conducted as needed.

Specific Study Aims and Methods

Aim 1: To evaluate Clinical Outcome Assessments (COAs) currently being used in premanifest HD. In accordance with the FDA, all types of COAs (a) Clinician-reported; (b) Observer-reported; (c) Patient-reported; and (d) Performance-based outcomes will be evaluated as appropriate for each phenotypic domain (motor, cognitive, psychiatric/behavioral, functional activity, quality of life). Specific outcomes of this aim will follow those recommended by the FDA including:

* a) Cross-sectional evaluation (critical for sample selection) of currently used COA instruments according to the following recommended criteria: mode of administration; format and scoring criteria; content validity; internal consistency reliability; test-retest reliability; floor and ceiling effects; construct validity; convergent validity; and strength of each COA expressed in terms of effect sizes.
* b) Longitudinal evaluation (critical for endpoint selection and responsiveness) of each COA to detect change using effect sizes across the premanifest and early HD disease continuum with documentation of the responder definition(s) of construct validity.
* c) Identification and documentation of the context of use (COU) and concept of interest (COI) for clinical trials in premanifest HD to position available COAs within a preliminary conceptual model.

Aim 2: To assess the psychometric properties of various biomarkers obtained from cerebral spinal fluid when compared between groups (premanifest HD, HD, NC) and over time (baseline and 2 years). Specific outcomes of this aim will include:

* a) CSF mHTT collected at baseline and 2 years in 100 premanifest HD, 25 diagnosed HD, and 25 healthy controls (HC) will be analyzed (blind to gene status) by two independent labs. Safety, feasibility, cost efficiency, and inter-site reliability will be obtained.
* b) Validity of CSF mutant huntingtin (mHTT) will be examined in HD groups for association with cross-sectional and longitudinal (a) phenotypic severity and decline using measures of the primary triad of clinical manifestation and progression (motor, cognitive, psychiatric/behavioral); (b) meaningful clinical outcome measures such as diagnosis in premanifest subjects and patient-reported outcomes, functional capacity and disability in all HD patients; and (c) available disease burden measures calculated as the product of Cytosine-Adenine-Guanine (CAG) repeat length and current age (considered a reflection of genetic toxicity by time survived; AKA disease burden). The investigators hypothesize that the candidate biomarkers will show appropriate association reflecting concurrent and predictive validity (types of criterion-related validity) with the most widespread "benchmarks" of HD phenotype, the Unified HD Rating Scale in diagnosed and advanced prodromal HD. Data from this Aim will immediately inform the interpretation of ongoing clinical trials that show biomarker levels in "some", but not "all", premanifest. Although it is unknown whether the biomarkers will demonstrate any predictive validity or concurrent validity for the entire premanifest HD group, data will immediately be useful to develop an evidence threshold for when in the premanifest HD prodrome, the biomarker will be detectable and tracked over time. The evidence threshold is immediately useful to the design of disease modifying trials in HD, particularly when the paramount goal is to prevent diagnosis, or manifestation.
* c) Biological criterion-related validity for biomarkers will be examined in HD groups for association with (a) microglial biomarkers; (b) inflammatory biomarkers; (c) neuronal death biomarkers; and (d) mHTT HD-specific protein. The investigators hypothesize that mHTT will show detection at the earliest point in the prodrome, followed by microglial markers, then inflammatory markers and, finally, neuron death markers in diagnosed HD.

ELIGIBILITY:
Inclusion Criteria for HD Participants:

* Estimated at low or high probability of motor diagnosis based on the multivariate risk score (MRS)
* Willing to commit to two in-person assessment visits (baseline and 2-year follow-up) and remote assessments as needed
* No active comorbidities (i.e. receiving stable treatment)
* All medications will be allowed although the protocol will mandate documentation of medications and analyses will particularly assess potential impact of medications on outcomes (i.e., sedation of abnormal movements)
* If previously measured, CAG results must be 36 or above (previous CAG is not a requirement, but this threshold will be upheld for those participants who have their CAG scores and/or have them in their medical record).

Inclusion Criteria for Healthy Controls (HC):

* Willing to commit to two in-person assessment visits (baseline and 2-year follow-up) and remote assessments as needed
* In generally good health
* IQ > 70
* Able to undergo an MRI scan

Exclusion Criteria (for all Participants):

* Evidence of unstable medical or psychiatric illness (including substance abuse)
* History of severe learning disability, mental retardation, or other central nervous system (CNS) disease or event (e.g., seizures, head trauma, additional neurological diagnoses)
* Treatment with phenothiazine-derivative antiemetic medications such as prochlorperazine, metoclopramide, promethazine and Inapsine greater than 3 times per month
* History of serious alcohol or drug abuse within the past year
* Unable (determined by patient's prescribing doctor) to not take tryptophan, leucine, niacin or niacinamide-containing dietary supplements, anti-inflammatory medications, anti-coagulants (such as warfarin and heparin) or anti-platelets (such as aspirin) in the past 14 days to assure safety during lumbar puncture
* Unable to fast (no food or drink, only water) overnight before the lumbar puncture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At baseline 258 male and female participants between the ages of 18 and 80 years will be enrolled in the study. Of the 258: 52 will be low risk of motor diagnosis, 102 high risk of motor diagnosis, 52 with diagnosed HD (stages I or II), and 52 age-, ethnicity-, and education-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Level | baseline
  UHDRS Motor Diagnosis of HD Diagnostic Confidence Level is a clinical rating of how confident the movement disorder specialist is that the person has manifest HD with over 99% confidence; scale is 0-4 where 0 is 'normal' and 4 is the highest motor dysfunction.
Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Level | 1 years
  UHDRS Motor Diagnosis of HD Diagnostic Confidence Level is a clinical rating of how confident the movement disorder specialist is that the person has manifest HD with over 99% confidence; scale is 0-4 where 0 is 'normal' and 4 is the highest motor dysfunction.
Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Level | 2 years
  UHDRS Motor Diagnosis of HD Diagnostic Confidence Level is a clinical rating of how confident the movement disorder specialist is that the person has manifest HD with over 99% confidence; scale is 0-4 where 0 is 'normal' and 4 is the highest motor dysfunction.
Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score | baseline
  UHDRS Total Motor Score is a 31-item instrument each item scored on a scale of 0-4 where 0 is 'normal' and 4 is the highest motor dysfunction. Total possible range of scores is 0-124.
Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score | 1 year
  UHDRS Total Motor Score is a 31-item instrument each item scored on a scale of 0-4 where 0 is 'normal' and 4 is the highest motor dysfunction. Total possible range of scores is 0-124.
Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score | 2 years
  UHDRS Total Motor Score is a 31-item instrument each item scored on a scale of 0-4 where 0 is 'normal' and 4 is the highest motor dysfunction. Total possible range of scores is 0-124.
Unified Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity | baseline
  UHDRS Total Functional Capacity is a clinician-rating scale of independence in activities of daily living. 13 is fully functioning and any drop in points in noted during pre-diagnosed HD.
Unified Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity | 1 year
  UHDRS Total Functional Capacity is a clinician-rating scale of independence in activities of daily living. 13 is fully functioning and any drop in points in noted during pre-diagnosed HD.
Unified Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity | 2 years
  UHDRS Total Functional Capacity is a clinician-rating scale of independence in activities of daily living. 13 is fully functioning and any drop in points in noted during pre-diagnosed HD.

SECONDARY OUTCOMES:
CANTAB composite score | baseline, 1 year, 2 years
  The Cambridge automated neuropsychological test battery (CANTAB) has a range of scores and will be summed across tasks for a composite. Higher scores will indicate better cognitive processing.
Cognitive Assessment Battery (CAB) Composite Score | baseline, 1 year, 2 years
  The CAB has a range of scores with higher scores indicative of better cognitive functions and a summed composite of the battery will be used as an outcome.
Tablet Cognitive Assessment Total (TabCat) Score | baseline, 1 year, 2 years
  The TabCat scores range across multiple tasks and the outcome will be a summed composite score across all cognitive tasks. Higher scores will indicate better cognitive processing.
Problem Behavior Assessment - short form (PBA) Score | baseline, 1 year, 2 years
  The PBA is an 11-item semi-structured instrument to assess the frequency and severity of behavioral symptoms of HD. Higher scores indicate increased severity and frequency of symptoms.

OTHER OUTCOMES:
Exploratory Measure: Cerebral Spinal Fluid Biomarker (BM) Assessment | baseline, 1 year, 2 years
  CSF will be processed at external labs for potential biomarkers of abnormality. CSF will be analyzed for Neurofilament light and mutant HTT.
Imaging BM measured via MRI | baseline, 1 year, 2 years
  MRI Biomarker will be the standardized volume of the basal ganglia.

CONTACTS AND LOCATIONS:
Overall Officials: Jane S Paulsen, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All clinical research data collected as part of this study is also stored in the NIH database for genotype and phenotypes (dbGaP) and the NIH National Data Archives for sharing with approved researchers worldwide. dbGaP provides two levels of access - open and controlled - in order to allow broad release of non-sensitive data, while providing oversight and investigator accountability for sensitive data sets involving personal health information. Summaries of studies and the contents of measured variables as well as original study document text are generally available to the public, while access to individual-level data including phenotypic data tables and genotypes require varying levels of authorization.
Supporting Information: Study Protocol
Time Frame: conclusion of study
Access Criteria: institutional certificate of professional degree

DOCUMENTS (1):
  • Informed Consent Form (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT04818060/ICF_000.pdf